CLINICAL TRIAL: NCT01729325
Title: Prevention of Post-Traumatic Stress Disorder in Relation to Appetitive Aggression in Burundian Soldiers Deployed in a Peace-keeping Mission in Somalia
Brief Title: Prevention of Post-Traumatic Stress Disorder in Soldiers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: The Volkswagen Foundation (Other)
Responsible Party: Principal Investigator, Anselm Crombach, Dipl.-Psych., University of Konstanz
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: UKULBUSO2012
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Post-traumatic Stress Disorder (PTSD); Aggressive Behavior
Keywords: Post-traumatic Stress disorder (PTSD); Aggressive Behavior; Appetitive Aggression; Resilience; Preventive Narrative Exposure Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Aggression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preventive Narrative Exposure Therapy (Experimental): Treatment with Pre-NET before deployment in peace-keeping mission
  Interventions: Behavioral: Preventive Narrative Exposure Therapy
- No treatment control (No Intervention)

INTERVENTIONS:
Behavioral: Preventive Narrative Exposure Therapy — During Pre-NET the client, with the assistance of the therapist, constructs a chronological narrative of his whole life with a focus on exposure to traumatic stress. Empathic understanding, active listening, congruency and unconditional positive regard are key components of the therapist's behavior who asks in detail for emotions, cognitions, sensory information, and physiological reactions, linking them to an autobiographical context. During two sessions a chronological overview of the whole life with a focus on traumatic events is developed and the most important traumatic experiences are processed.
  Arms: Preventive Narrative Exposure Therapy

SUMMARY:
Soldiers in conflict or former conflict regions deployed in peace-keeping missions were and are often exposed to multiple traumatic events and situations in which they are forced to engage in violent behavior. The Preventive Narrative Exposure Therapy (Pre-NET) aims to reinforce resilience thereby reducing the risk of developing or aggravating PTSD or other mental disorders as a result of traumatic experiences. The effective prevention of mental disorders as a result of war deployment is expected to facilitate reintegration in civil life after deployment and reduce uncontrolled violence.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to traumatic experiences derived from expert interviews with scores of the Traumatic Life Event List for War and Torture
* Soldiers are part of the Burundian army and of the joint African Union and United Nations peacekeeping mission in Somalia (AMISOM)

Exclusion Criteria:

* Current use of mind altering drugs
* Psychotic symptoms

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Severity of traumatic symptoms measured via the Post-traumatic Stress Disorder Scale-Interview (PSS-I) | 15 months
Extend of appetitive aggression via the Appetitive Aggressions Scale (AAS) | 15 months

SECONDARY OUTCOMES:
Severity of depressive symptoms measured via the Patient Health Questionnaire-9 (PHQ-9) | 15 months
Strength of suicidal ideation measured via the MINI | 15 months
Physical health complains | 15 months

CONTACTS AND LOCATIONS:
Locations (1):
- Burundian Army (FDN), Bujumbura, Bujumbura Mairie Province, Burundi